CLINICAL TRIAL: NCT01911871
Title: Multicenter Observational Study on Myocardial Iron Overload in 3 Multitransfused Populations
Acronym: SUFEMYO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI10071; RAF11005
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Thalassemia; Sickle Cell Disease; Myelodysplasia
Keywords: Thalassemia; sickle cell disease; myelodysplasia; transfusion; chelation
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell; Anemia, Refractory, with Excess of Blasts | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- thalassemia: patients affected with thalassemia
  Interventions: Biological: Blood sample
- sickle cell disease: patients affected with sickle cell disease
  Interventions: Biological: Blood sample
- myelodysplasia: patients affected with myelodysplasia
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — a blood sample was taken on the day of inclusion

SUMMARY:
The investigators' primary objective is to study prevalences of myocardial iron overload, defined as a cardiac T2*< 20 ms, in 3 populations of multiply transfused patients, affected with thalassemia, sickle cell disease, and myelodysplasia.

DETAILED DESCRIPTION:
The inevestigators' primary objective is to study prevalences of myocardial iron overload, defined as a cardiac T2*< 20 ms, in 3 populations of multiply transfused patients, affected with thalassemia, sickle cell disease, and myelodysplasia.

The investigators will record concomitantly parameters which, according to literature data, may influence the occurrence of this complication, and will look for correlations with these parameters and iron overload (secondary objectives), in each of the 3 cohorts.

14 centres are involved and enrol patients with thalassemia, or sickle cell disease, or myelodysplasia having received in the past year > 8 erythrocyte concentrates, and having had a cardiac MRI. Patients files register the type of the disease, age at the beginning of transfusion and chelation, chelator type and dosage, liver and cardiac T2*.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia, sickle cell disease, myelodysplasia
* having received in the past year > 8 erythrocyte concentrates
* > 6 years of age

Exclusion Criteria:

* preexisting cardiac disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients affected with thalassemia, SCD, and myelodysplasia
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cardiac T2* (MRI) | Day 0

SECONDARY OUTCOMES:
Liver T2*(MRI) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Mariane de montalembert, MD/PhD, Study Director — Groupement Hospitalier Necker
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Result] de Montalembert M, Ribeil JA, Brousse V, Guerci-Bresler A, Stamatoullas A, Vannier JP, Dumesnil C, Lahary A, Touati M, Bouabdallah K, Cavazzana M, Chauzit E, Baptiste A, Lefebvre T, Puy H, Elie C, Karim Z, Ernst O, Rose C. Cardiac iron overload in chronically transfused patients with thalassemia, sickle cell anemia, or myelodysplastic syndrome. PLoS One. 2017 Mar 3;12(3):e0172147. doi: 10.1371/journal.pone.0172147. eCollection 2017. PMID 28257476